CLINICAL TRIAL: NCT05166057
Title: Telerehabilitation in Patients With Fibrosing Interstitial Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, ESRA PEHLIVAN, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLD_Tele
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Fibrosing Interstitial Lung Disease; Telerehabilitation
Keywords: fibrosing interstitial lung disease; telerehabilitation; physiotherapy; pulmonary rehabilitation

STUDY DESIGN:
Intervention Model Description: The cases meeting the inclusion criteria will be randomized and divided into three groups, the groups will be named as Telerehabilitation Exercise Group (TGr), Video Group (VGr) and Standard pulmonary rehabilitation group (SGr).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation Group (TG) (Experimental): TGr will be given online exercises, synchronized 2 days a week, and a home program for 1 day, accompanied by a physiotherapist, via videoconference on the group smartphone.
  Interventions: Other: Synchronized online telerehabilitation exercise program
- Video Group (VGr) (Experimental): After 1 session of online simultaneous exercise training in the company of a physiotherapist via a smart phone videoconference to the VGr group, an exercise video including the exercises will be sent and the participants will be asked to do exercises 3 days a week. The cases will be asked to keep an exercise diary and the status of the diaries will be followed by calling once a week.
  Interventions: Other: Videobased telerehabilitation exercise program
- Standard pulmonary rehabilitation group (SGr) (Experimental): The SGr group will be applied the pulmonary rehabilitation program with supervision in the hospital 2 days a week, and participants will be asked to do exercises at home for 1 day. The exercise period will be 8 weeks for both groups.
  Interventions: Other: Hospital based outpatient exercise program

INTERVENTIONS:
Other: Synchronized online telerehabilitation exercise program — Breathing exercises, inspiratory muscle training, peripheral muscle strengthening training and gait training will be applied to the patient by videoconference.
  Arms: Telerehabilitation Group (TG)
Other: Videobased telerehabilitation exercise program — A video containing breathing exercises, inspiratory muscle training, peripheral muscle strengthening training and gait training will be given to the patient and will be asked to exercise regularly.
  Arms: Video Group (VGr)
Other: Hospital based outpatient exercise program — Breathing exercises, inspiratory muscle training, peripheral muscle strengthening training and gait training will be applied to the patient in the hospital..
  Arms: Standard pulmonary rehabilitation group (SGr)

SUMMARY:
The aim of the study is to determine the effectiveness of different exercise programs applied to 3 groups randomly formed in patients with fibrosing interstitial lung disease (FILD).

Secondary purpose: To determine the feasibility and effectiveness of telerehabilitation in FILD cases.

DETAILED DESCRIPTION:
The cases meeting the inclusion criteria will be randomized and divided into three groups, the groups will be named as Telerehabilitation Exercise Group (TGr), Video Group (VGr) and Standard pulmonary rehabilitation group (SGr).TGr will be given online exercises, synchronized 2 days a week, and a home program for 1 day, accompanied by a physiotherapist, via videoconference on the group smartphone.After 1 session of online simultaneous exercise training in the company of a physiotherapist via a smart phone videoconference to the VGr group, an exercise video including the exercises will be sent to participants and the patients will be asked to do exercises 3 days a week. The participants will be asked to keep an exercise diary and the status of the diaries will be followed by phone call once a week.The SGr group will be applied the pulmonary rehabilitation program with supervision in the hospital 2 days a week, and participants will be asked to do exercises at home for 1 day. The exercise period will be 8 weeks for both groups.Details of the exercises to be applied to the cases are as follows: The exercise program includes aerobic, resistance exercises and breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* Have a diagnosis of fibrosing interstitial lung disease diagnosed according to the clinical diagnostic criteria of the American Thoracic and European Respiratory Societies (ATS-ERS).
* Presence of dyspnea on exertion Stable clinical state at the time of admission without infection or exacerbation in the previous 4 weeks
* Ability to use a smart phone

Exclusion Criteria:

* Patients with severe comorbid diseases, unstable coronary artery disease, collagen vascular diseases and needing high flow oxygen therapy (˃ 3-4 L \min).
* history of effort-related syncope or any comorbidity (such as severe orthopedic or neurological deficits or unstable heart disease) that precludes exercise training.
* Participating in a pulmonary rehabilitation program within the past 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2022-01-22 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | Change from baseline at 2 months
  The 6-minute walking test will conduct in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Participants will ask to walk as far as they can. Prior to and following the test, oxygen saturation, heart rate and Borg fatigue rating will measure, and the walking distance will record.
Dyspnea perception | Change from baseline at 2 months
  modified Medical Council Dyspnea score will rate the sensation of dyspnea as the person perceives it.The severity of dyspnea is rated on a scale of 0 to 4."0 point" means no dyspnea perception and "4point" means severe dyspnea perception.
Fatigue severity | Change from baseline at 2 months
  The fatigue severity scale: A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity.
  The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity Another way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7 Self-report scale

SECONDARY OUTCOMES:
Respiratory muscle strength | Change from baseline at 2 months
  The mouth pressure measurement (maximum inspiratory and expiratory pressure) will perform with the Pony Fx spirometry device. Patient will place a rubber mouthpiece with flanges, on the device, exhale/inhale slowly and completely, and then will try to breath in as hard as possible. The patient will allow to rest for about a minute and the maneuver will repeat. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value will obtain.
Physical activity level | Change from baseline at 2 months
  The International Physical Activity Questionnaire (IPAQ) was developed as an instrument for cross-national monitoring of physical activity and inactivity. This measure assesses the types of intensity of physical activity and sitting time that people do as part of daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Anxiety level | Change from baseline at 2 months
  Hospital Anxiety Depression scale:The levels of anxiety will asses by Hospital Anxiety Depression Scale (HADS) .The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).Several studies suggest a cut-off score of ≥8 to be optimal for best sensitivity and specificity. The HADS has sensitivity and specificity of about 80%, and a predictive validity for identification of about 70%.
Depression level | Change from baseline at 2 months
  Hospital Anxiety Depression scale:The levels of depression will asses by Hospital Anxiety Depression Scale (HADS) .The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).Several studies suggest a cut-off score of ≥8 to be optimal for best sensitivity and specificity. The HADS has sensitivity and specificity of about 80%, and a predictive validity for identification of about 70%.
Quality of life level | Change from baseline at 2 months
  Saint George Respiratory Questionaire (SGRQ) score: The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Pulmonary function tests (PFTs) | Change from baseline at 2 months
  PFTs will perform by using the Pony Fx spirometry device, and according to the American Thoracic Society (ATS) guidelines

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Pehlivan, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pehlivan E, Cetinkaya E, Karaahmetoglu FS, Ozcan ZB, Baydili KN, Demirkol B, Cinarka H, Eren R, Atac A. The impact of different pulmonary rehabilitation approaches on fibrotic interstitial lung disease: a comparative randomized trial. Expert Rev Respir Med. 2025 Sep;19(9):1027-1035. doi: 10.1080/17476348.2025.2513512. Epub 2025 May 29. PMID 40440705